CLINICAL TRIAL: NCT02584309
Title: A Non-Inferiority Study of Doxorubicin With Upfront Dexrazoxane for the Treatment of Advanced or Metastatic Soft Tissue Sarcoma
Brief Title: Doxorubicin With Upfront Dexrazoxane for the Treatment of Advanced or Metastatic Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201510049
Record Dates: First submitted 2015-10-12; First posted 2015-10-22 (Estimated); Results first posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Sarcoma, Soft Tissue; Soft Tissue Sarcoma; Undifferentiated Pleomorphic Sarcoma; Leiomyosarcoma; Liposarcoma; Synovial Sarcoma; Myxofibrosarcoma; Angiosarcoma; Fibrosarcoma; Malignant Peripheral Nerve Sheath Tumor; Epithelioid Sarcoma
MeSH Terms: conditions — Sarcoma; Histiocytoma, Malignant Fibrous; Leiomyosarcoma; Liposarcoma; Sarcoma, Synovial; Dermatofibrosarcoma; Hemangiosarcoma; Fibrosarcoma; Neurofibrosarcoma | interventions — Dexrazoxane; Razoxane; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Doxorubicin and Upfront Dexrazoxane (Experimental): * Dexrazoxane will be given intravenously on an outpatient basis over 15 minutes on each day that doxorubicin is given.
  * Dexrazoxane should be given no more than 30 minutes prior to administration of doxorubicin, which is typically given on Day 1 of a 21-day cycle.
  * Dosing is a 10:1 ratio of dexrazoxane to doxorubicin; doxorubicin is typically given at 75 mg/m2, so dexrazoxane dosing would be 750 mg/m2.
  * In the event of a national shortage of dexrazoxane, 72-hour infusional doxorubicin can be used instead of dexrazoxane and bolus doxorubicin..
  Interventions: Drug: Dexrazoxane; Drug: Doxorubicin
- Arm 2: control (Doxorubicin and Standard of Care Dexrazoxane) (Active Comparator): * Doxorubicin is given as standard of care. Doxorubicin is typically given at 75 mg/m2 on Day 1 of a 21-day cycle.
  * Starting with cycle 5, standard of care dexrazoxane (75 mg/m2) will be given for 4 cycles.
  * The last 10 patients enrolled after completion of enrollment to Arm 1 will be enrolled to Arm 2.
  Interventions: Drug: Dexrazoxane; Drug: Doxorubicin

INTERVENTIONS:
Drug: Dexrazoxane
  Other Names: Zinecard®; Totect®
Drug: Doxorubicin
  Other Names: Adriamycin; Hydroxydaunomycin Hydrochloride; Hydroxydoxorubicin Hydrochloride; Rubex

SUMMARY:
The purpose of this research study is to look at whether giving a drug called dexrazoxane with standard of care doxorubicin affects the progression of the disease. Dexrazoxane is often given at the same time as doxorubicin to help reduce the incidence and severity of disease of the heart muscle (which can be caused by doxorubicin).

In January 2019 Eli Lilly and Company reported that the results of the Phase 3 study of olaratumab (Lartruvo), in combination with doxorubicin in patients with advanced or metastatic soft tissue sarcoma, did not confirm the clinical benefit of olaratumab in combination with doxorubicin as compared to doxorubicin alone. Therefore olaratumab is being removed from the front line standard of care regimen. Amendment #9 was made to the protocol to reflect these changes to the standard of care treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed grade 2 or 3 soft tissue sarcoma that is unresectable or metastatic. Surgery for primary or metastatic disease after chemotherapy following a response is allowed. Patients with the following tumor types are eligible:

  * Undifferentiated pleomorphic sarcoma
  * Leiomyosarcoma
  * Malignant fibrous histiocytoma
  * Liposarcoma (myxoid/round cell, pleomorphic or dedifferentiated)
  * Synovial sarcoma
  * Myxofibrosarcoma
  * Angiosarcoma
  * Fibrosarcoma
  * Malignant peripheral nerve sheath tumor
  * Epithelioid sarcoma
  * Unclassified high-grade sarcoma (not otherwise specified)
  * Soft tissue sarcoma for which treatment with an anthracycline is appropriate at the approval of the Principal Investigator (PI)
* Measurable disease according to RECIST 1.1; that is, measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm with CT scan, as ≥ 20 mm by chest x-ray, or ≥ 10 mm with calipers by clinical exam.
* Planning to initiate treatment with doxorubicin (starting dose 75 mg/m2) as routine care.
* Prior adjuvant chemotherapy with gemcitabine and/or docetaxel/paclitaxel is allowed.
* At least 18 years of age.
* ECOG performance status of 0 or 1
* Adequate organ function defined as:

  * Leukocytes ≥ 3,000/mcL
  * Absolute neutrophil count ≥ 1,500/mcl
  * Platelets ≥ 100,000/mcl
  * Total bilirubin ≤ 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
  * Creatinine ≤ IULN OR Creatinine clearance ≥ 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal. Creatinine clearance should be calculated using the actual weight from day 1 of cycle
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Able to understand and willing to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Myocardial infarction within the past 12 months, or stable or unstable angina.
* Systolic heart failure defined as left ventricular ejection fraction ≤ 45%.
* Symptomatic valvular heart disease.
* Prior chemotherapy for advanced or metastatic disease.
* Known brain metastases.
* Prior or second primary malignancies within the last two years (except carcinoma in situ of the cervix, non-metastatic prostate cancer, or basal cell or squamous cell carcinoma of the skin which were treated with local resection only; prior adjuvant androgen deprivation therapy in the case of prostate cancer is permitted, but current adjuvant androgen deprivation therapy is not).
* Currently receiving any investigational agents.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to dexrazoxane or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and/or breastfeeding. Patient must have a negative pregnancy test within 14 days of study entry.
* Known HIV-positivity on combination antiretroviral therapy because of the potential for pharmacokinetic interactions with dexrazoxane. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Prior treatment with anthracyclines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2016-02-22 (Actual); Primary Completion 2022-07-17 (Actual); Study Completion 2022-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian A Van Tine, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Unassigned Arm: The participant was enrolled but withdrew prior to starting treatment.
Period: Overall Study
Arm/Group | Arm 1: Doxorubicin and Upfront Dexrazoxane | Arm 2: Control (Doxorubicin and Standard of Care Dexrazoxane) | Unassigned Arm
Started | 62 | 10 | 1
Completed | 62 | 10 | 0
Not Completed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Doxorubicin and Upfront Dexrazoxane | Arm 2: Control (Doxorubicin and Standard of Care Dexrazoxane) | Unassigned Arm | Total
Number analyzed (Participants) | 62 | 10 | 1 | 73
Age, Continuous [Median (Full Range); unit: years] | 65 [23 to 85] | 62.5 [55 to 71] | 54 [54 to 54] | 65 [23 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 5 | 0 | 38
  Male | 29 | 5 | 1 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 61 | 10 | 1 | 72
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 0 | 0 | 8
  White | 54 | 10 | 1 | 65
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 62 | 10 | 1 | 73

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) (Arm 1 Only)
Description: * PFS is defined as the time from on study to the first occurrence of progression or death, whichever occurs first.
  * If no event exists, the PFS will be censored at the last follow-up.
  * Progressive disease - At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
Time Frame: Up to 5 years
Population: Participants enrolled in Arm 2 are not evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1: Doxorubicin and Upfront Dexrazoxane | Arm 2: Control (Doxorubicin and Standard of Care Dexrazoxane)
Number analyzed (Participants) | 62 | 0
months | 5.48 [4.01 to 7.37] |

2. Secondary Outcome: Cardiac-related Mortality
Description: Death due to cardiovascular while on study (heart failure, myocardial infarction, fatal arrhythmia).
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Doxorubicin and Upfront Dexrazoxane | Arm 2: Control (Doxorubicin and Standard of Care Dexrazoxane)
Number analyzed (Participants) | 62 | 10
Participants | 0 | 0

3. Secondary Outcome: Percentage of Patients With Heart Failure or Cardiomyopathy
Description: * Cardiomyopathy is now referred to as cancer therapy related cardiac dysfunction (CTRCD) by the recent consensus statement of the International Cardio-Oncology Society. Moderate CTRCD is defined as >10% ejection fraction drop to <50%. Mild CTRCD is defined as drop in ≥15% ventricular strain or if no ventricular strain, a drop in ejection fraction of ≥50%.
  * Heart failure is defined according to the recent Universal Definition and Classification of Heart Failure: A Report of the Heart Failure Society of America, Heart Failure Association of the European Society of Cardiology, Japanese Heart Failure Society and Writing Committee of the Universal Definition of Heart Failure.
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Doxorubicin and Upfront Dexrazoxane | Arm 2: Control (Doxorubicin and Standard of Care Dexrazoxane)
Number analyzed (Participants) | 62 | 10
Participants
  Moderate cancer therapy related cardiac dysfunction (CTRCD) | 4 | 0
  Mild cancer therapy related cardiac dysfunction (CTRCD) | 25 | 4
  Heart failure with mildly reduced ejection fraction (HfmrEF) | 0 | 0
  Heart failure with preserved ejection fraction (HFpEF) | 17 | 1

4. Secondary Outcome: Ability of 3D Echocardiogram to Serve as an Early Marker of Cardiac Dysfunction Compared to 2D Echocardiogram Modified Simpson's Biplane Method of LVEF
Description: * Cardiac dysfunction for this outcome measure is defined as moderate cancer therapy related cardiac dysfunction (CTRCD) as assessed by 2D Echocardiogram Modified Simpson's Biplane Method of LVEF. Moderate CTRCD is defined as >10% ejection fraction drop to <50%.
  * 3D echocardiograms were reviewed for evidence of cardiac dysfunction prior to onset of Moderate CTRCD by 2D echocardiogram. Dysfunction on 3D Echo was defined as >10% ejection fraction drop to <50%.
Time Frame: Baseline and day 1 of each odd numbered cycle (each cycle is 21 days) up to 1 year
Population: 13 participants were removed due to lack of analyzable 3D echo prior to onset of Moderate CTRCD or end of study.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Doxorubicin and Upfront Dexrazoxane | Arm 2: Control (Doxorubicin and Standard of Care Dexrazoxane)
Number analyzed (Participants) | 46 | 9
Participants
  Patients with moderate CTRCD by 2D echo: number analyzed (Participants) | 1 | 0
  Patients with moderate CTRCD by 2D echo: Early dysfunction noted on 3D Echo | 0 | 0
  Patients with moderate CTRCD by 2D echo: No early dysfunction noted on 3D echo | 1 | 0
  Patients without moderate CTRCD by 2D echo: number analyzed (Participants) | 45 | 9
  Patients without moderate CTRCD by 2D echo: Early dysfunction noted on 3D Echo | 7 | 0
  Patients without moderate CTRCD by 2D echo: No early dysfunction noted on 3D echo | 38 | 9

5. Secondary Outcome: Early Detection of Cardiac Dysfunction by 2D Echocardiography Ventricular Strain Compared to 2D Echocardiography Ejection Fraction
Description: * Cardiac dysfunction for this outcome measure is defined as moderate cancer therapy related cardiac dysfunction (CTRCD) by 2D Echocardiogram Modified Simpson's Biplane Method of LVEF. Moderate CTRCD is defined as >10% ejection fraction drop to <50%.
  * Patients were assessed for early evidence of dysfunction by strain defined as a relative drop in global longitudinal strain (GLS) by 15% and GLS > -17%.
Time Frame: Baseline and day 1 of each odd numbered cycle (each cycle is 21 days) up to 1 year
Population: Participants were not included in this outcome measure if they did not have GLS.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Doxorubicin and Upfront Dexrazoxane | Arm 2: Control (Doxorubicin and Standard of Care Dexrazoxane)
Number analyzed (Participants) | 48 | 10
Participants
  Patients with moderate CTRCD by 2D echo: number analyzed (Participants) | 2 | 0
  Patients with moderate CTRCD by 2D echo: Early dysfunction noted on 2D GLS | 1 | 0
  Patients with moderate CTRCD by 2D echo: No early dysfunction noted on 2D GLS | 1 | 0
  Patients without moderate CTRCD by 2D echo: number analyzed (Participants) | 46 | 10
  Patients without moderate CTRCD by 2D echo: Early dysfunction noted on 2D GLS | 6 | 2
  Patients without moderate CTRCD by 2D echo: No early dysfunction noted on 2D GLS | 40 | 8

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of treatment through 30 days following last day of treatment. The median follow-up was 142 days (full range 9-1214 days). All-cause mortality was collected from start of treatment through completion of follow-up. The median follow-up was 529 days (full range 9-2188 days).
Arm/Group | Arm 1: Doxorubicin and Upfront Dexrazoxane | Arm 2: Control (Doxorubicin and Standard of Care Dexrazoxane)
All-Cause Mortality (participants affected / at risk) | 52/62 | 5/10
Serious Adverse Events (participants affected / at risk) | 17/62 | 1/10
Other Adverse Events (participants affected / at risk) | 62/62 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Doxorubicin and Upfront Dexrazoxane (N=62) | Arm 2: Control (Doxorubicin and Standard of Care Dexrazoxane) (N=10)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Fever (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Sudden death NOS (General disorders) | 1 | 0
Sepsis (Infections and infestations) | 3 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 0
Suicide (Psychiatric disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Doxorubicin and Upfront Dexrazoxane (N=62) | Arm 2: Control (Doxorubicin and Standard of Care Dexrazoxane) (N=10)
Anemia (Blood and lymphatic system disorders) | 58 | 10
Febrile neutropenia (Blood and lymphatic system disorders) | 19 | 3
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 1 | 0
Myositis (Cardiac disorders) | 1 | 0
Non-cardiac chest pain (Cardiac disorders) | 3 | 0
Palpitations (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0
Ear sensitivity (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Hyperparathyroidism (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 2 | 0
Blurred vision (Eye disorders) | 4 | 0
Glaucoma (Eye disorders) | 1 | 0
Watering eyes (Eye disorders) | 3 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 10 | 1
Anal hemorrhage (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 2 | 0
Bleeding hemorrhoids (Gastrointestinal disorders) | 1 | 0
Bloating (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 31 | 6
Diarrhea (Gastrointestinal disorders) | 17 | 3
Dry mouth (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 4 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 | 0
Gum bleeding (Gastrointestinal disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 2 | 0
Lip swelling (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 20 | 3
Nausea (Gastrointestinal disorders) | 24 | 8
Oral dysethesia (Gastrointestinal disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 3 | 0
Rectal bleeding (Gastrointestinal disorders) | 1 | 0
Rectal ulcer (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Stomach pain (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 15 | 1
Chills (General disorders) | 6 | 0
Edema limbs (General disorders) | 27 | 1
Edema trunk (General disorders) | 2 | 0
Fatigue (General disorders) | 49 | 7
Fever (General disorders) | 18 | 2
Flu like symptoms (General disorders) | 4 | 1
Infusion-related reaction (General disorders) | 8 | 0
Localized edema (General disorders) | 1 | 0
Malaise (General disorders) | 4 | 0
Pain (General disorders) | 1 | 0
Allergic reaction (Immune system disorders) | 1 | 0
Bacteremia (Infections and infestations) | 1 | 0
Eye infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 5 | 1
Mucosal infection (Infections and infestations) | 1 | 0
Nail infection (Infections and infestations) | 2 | 0
Papulopastular rash (Infections and infestations) | 3 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Rash pustular (Infections and infestations) | 1 | 1
Rhinitis infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 4 | 0
Sinusitis (Infections and infestations) | 3 | 0
Skin infection (Infections and infestations) | 2 | 0
Tooth infection (Infections and infestations) | 1 | 0
Upper respiratory infection (Infections and infestations) | 5 | 0
Urinary tract infection (Infections and infestations) | 10 | 0
Vaginal infection (Infections and infestations) | 1 | 0
Wound complication (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 3 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 4 | 0
Activated partial thromboplastin time prolonged (Investigations) | 13 | 0
Alanine aminotransferase increased (Investigations) | 12 | 1
Alkaline phosphatase increased (Investigations) | 16 | 5
Aspartate aminotransferase increased (Investigations) | 13 | 0
Blood bilirubin increased (Investigations) | 4 | 0
Cholesterol high (Investigations) | 4 | 0
Creatinine increased (Investigations) | 6 | 5
Ejection fraction decreased (Investigations) | 7 | 0
GGT increased (Investigations) | 2 | 0
INR increased (Investigations) | 22 | 1
Lymphocytes decreased (Investigations) | 48 | 9
Neutrophil count decreased (Investigations) | 43 | 3
Platelet count decreased (Investigations) | 22 | 3
White blood cell decreased (Investigations) | 29 | 4
Anorexia (Metabolism and nutrition disorders) | 15 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Failure to thrive (Metabolism and nutrition disorders) | 2 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 14 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 4 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 1
Hypernatremia (Metabolism and nutrition disorders) | 11 | 3
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 33 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 26 | 7
Hypoglycemia (Metabolism and nutrition disorders) | 9 | 0
Hypokalemia (Metabolism and nutrition disorders) | 19 | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 4 | 0
Hyponatremia (Metabolism and nutrition disorders) | 24 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 8 | 3
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Knee pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle aches (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle pain (Musculoskeletal and connective tissue disorders) | 7 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 1
Neuroma (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 2
Pelvic pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Thigh pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 0
Akathisia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 4 | 0
Dysarthria (Nervous system disorders) | 2 | 0
Dysgeusia (Nervous system disorders) | 6 | 0
Dysphasia (Nervous system disorders) | 3 | 0
Extrapyramidal disorder (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 18 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 6 | 2
Phantom pain (Nervous system disorders) | 2 | 0
Sinus pain (Nervous system disorders) | 1 | 1
Spasticity (Nervous system disorders) | 4 | 1
Syncope (Nervous system disorders) | 3 | 0
Tremor (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 7 | 5
Confusion (Psychiatric disorders) | 3 | 0
Depression (Psychiatric disorders) | 2 | 1
Hallucinations (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 6 | 0
Irritability (Psychiatric disorders) | 1 | 0
Mental status altered (Psychiatric disorders) | 1 | 0
Psychosis (Psychiatric disorders) | 1 | 0
Restlessness (Psychiatric disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 14 | 1
Proteinuria (Renal and urinary disorders) | 9 | 1
Urinary frequency (Renal and urinary disorders) | 2 | 0
Elevated PSA (Reproductive system and breast disorders) | 1 | 0
Penile pain (Reproductive system and breast disorders) | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Post nasal drip (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 9 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 21 | 10
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0
Hand and foot syndrome (Skin and subcutaneous tissue disorders) | 2 | 0
Nail discoloration (Skin and subcutaneous tissue disorders) | 4 | 0
Nail loss (Skin and subcutaneous tissue disorders) | 2 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 4 | 0
Nodule left forearm (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Photosensitivity (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 0
Rash non pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Subcutaneous tissue disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Sweating (Skin and subcutaneous tissue disorders) | 1 | 0
Tick bites (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0
Capillary leak syndrome (Vascular disorders) | 1 | 0
Flushing (Vascular disorders) | 0 | 2
Hot flashes (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 8 | 0
Hypotension (Vascular disorders) | 5 | 1
Intercardial thrombic (Vascular disorders) | 1 | 0
Lymphedema (Vascular disorders) | 3 | 0
Superficial thrombophlebitis (Vascular disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 14 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT02584309/Prot_SAP_000.pdf